CLINICAL TRIAL: NCT03149666
Title: Anthropometric Variables and Perception of Bitter Taste in Obese Adults or Not
Brief Title: Quantitative Evaluation of Bitter Taste in Obesity
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Julio Sergio Marchini, Principal Investigator, University of Sao Paulo
Other Study IDs: HCRP 924/2015
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of bitter taste: Participants will be evaluated as to the intensity of bitter taste when performing watery mouthwash with quinine.

SUMMARY:
Although taste influences food choices and favours diseases like obesity, there is no consensus about the existence of correlations between bitterness and anthropometric variables. Also, an electronic-based method for data collection could provide a more appropriate way for the evaluation of taste perception and save time.

The objective is to search for correlations between bitterness and anthropometric variables.

DETAILED DESCRIPTION:
A cross-sectional study evaluating correlations between the bitterness rates given on a generalized Labeled Magnitude Scale, anthropometrics and other variables. Bitterness perceptions at the tip of the tongue (TOTp) and at the whole mouth (WMp) were recorded using a locally developed novel cloud-based software (Cloud-gLMS). The ANCOVA test was adjusted using TOTp and WMp as dependent variables and age, height, weight, BMI, gender, waist circumference, alcohol intake, comorbidities, and use of medications as independent variables.

ELIGIBILITY:
Inclusion Criteria:

* Weight limit of 150 kg and who are able to read the text with the guidelines on how to be punctuated the sensation of bitter in the generalized labeled scale.

Exclusion Criteria:

* Being a relative of the first degree of a patient already included in the research, tobacco in the forms of cigarettes, pipes and cigars in the last 30 days, presence of coryza, nasal congestion or frequent sneezing, dental treatment on the same day of the research. Being a dementia sufferer, having an altered, drowsy level of consciousness. Show upper limb tremor visible.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy people without obesity and people with obesity.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of bitter taste 1 | 1 time
  It will be gently applied at the end of the tongue, by means of a swab soaked in the quinine solution at room temperature, in continuous movements from left to right, and will point a note to the bitter level.
Sensitivity of bitter taste 2 | 1 time
  The volunteer will perform a "mouthwash" with the quinine solution, and will point a note to the bitter level.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reiter ER, DiNardo LJ, Costanzo RM. Toxic effects on gustatory function. Adv Otorhinolaryngol. 2006;63:265-277. doi: 10.1159/000093765. PMID 16733344
- [Background] Sharma K, Kaur GK. PTC bitter taste genetic polymorphism, food choices, physical growth in body height and body fat related traits among adolescent girls from Kangra Valley, Himachal Pradesh (India). Ann Hum Biol. 2014 Jan-Feb;41(1):29-39. doi: 10.3109/03014460.2013.822929. Epub 2013 Aug 12. PMID 23937293
- [Background] Keller KL, Adise S. Variation in the Ability to Taste Bitter Thiourea Compounds: Implications for Food Acceptance, Dietary Intake, and Obesity Risk in Children. Annu Rev Nutr. 2016 Jul 17;36:157-82. doi: 10.1146/annurev-nutr-071715-050916. Epub 2016 Apr 6. PMID 27070900
- [Background] Bartoshuk LM, Duffy VB, Green BG, Hoffman HJ, Ko CW, Lucchina LA, Marks LE, Snyder DJ, Weiffenbach JM. Valid across-group comparisons with labeled scales: the gLMS versus magnitude matching. Physiol Behav. 2004 Aug;82(1):109-14. doi: 10.1016/j.physbeh.2004.02.033. PMID 15234598
- [Background] Segovia C, Hutchinson I, Laing DG, Jinks AL. A quantitative study of fungiform papillae and taste pore density in adults and children. Brain Res Dev Brain Res. 2002 Oct 20;138(2):135-46. doi: 10.1016/s0165-3806(02)00463-7. PMID 12354641